CLINICAL TRIAL: NCT03475147
Title: Validation of a Smartphone-Based Flicker Fusion Test
Brief Title: Smartphone Flicker Fusion Test for Patients With Optic Disorders.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Randy Kardon (Other)
Responsible Party: Sponsor-Investigator, Randy Kardon, MD, PhD, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 201610703
Record Dates: First submitted 2018-03-16; First posted 2018-03-23 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-05

CONDITIONS: Scotoma
MeSH Terms: conditions — Scotoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- eyeFusion Control Subjects (Active Comparator): Healthy normal controls with no known eye disorders age 18-80.
  Interventions: Device: eyeFusion
- eyeFusion Patients (Experimental): Scotoma subjects aged 18-80.
  Interventions: Device: eyeFusion

INTERVENTIONS:
Device: eyeFusion — Smartphone app based flicker fusion test.

SUMMARY:
The purpose of this project is to validate a quick, easy-to-use and administer smartphone flicker fusion test. The app (called eyeFusion) can potentially be used to easily and quickly collect critical flicker fusion measurements on patients admitted with optic disorders as part of the clinical care process.

DETAILED DESCRIPTION:
The smartphone app developed is a flicker fusion that presents the subject with a series of stimuli consisting of a flickering pattern of bars above or below a static rectangle. For each stimulus presentation, the user has to tap the region that is flickering. The duration of the app is less than 2 minutes.

This study will assess the validity of the test construct in measuring flicker fusion thresholds, and serve as a foundation for further iterative designs of the app and future validation and characterization studies.

ELIGIBILITY:
Inclusion Criteria:

Control

* Age matched 18-80 years of age.
* Healthy normal controls with no known eye disorders.

Exclusion Criteria:

* Scotoma or any other ocular disorder

Inclusion Criteria - Patients

* Age 18-80
* Clinically associated scotoma

Exclusion Criteria - Patients

-Any other ocular disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-01-27 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Assess Validity of the test construct measuring flicker fusion thresholds. | 1/1/2020
  The smartphone app developed is a flicker fusion that presents the subject with a series of stimuli consisting of a flickering pattern of bars above or below a static rectangle. The study will assess the validity of the test construct in measuring flicker fusion thresholds, and serve as a foundation for further iterative designs of the app and future validation and characterization studies.

CONTACTS AND LOCATIONS:
Overall Officials: Randy Kardon, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No